CLINICAL TRIAL: NCT04575792
Title: Effect of Oral Habits on Orofacial Dysfunction and Oral Health Related Quality of Life Among a Group of Egyptian Children: Cohort Study
Brief Title: Oral Habits Effect on Orofacial Dysfunction and Oral Health Related Quality of Life.
Acronym: OHRQoL
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf Abd Elsabour Abd Elkareem, Principal Investigator, Cairo University
Other Study IDs: 1111
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Oral Habits; Oro-Facial Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C group: C group: control group, children who do not practice oral habits.
- E group: E group: exposed group, children who practicing oral habits.
  Interventions: Behavioral: Practicing oral habits

INTERVENTIONS:
Behavioral: Practicing oral habits — children who practice one or more of the specified oral habits ( mouth breathing, object sucking, or tongue thrusting) are considered exposed.
  Groups: E group

SUMMARY:
The aim of the present study is to determine the effect of oral habits on orofacial dysfunction and oral health related quality of life among a group of Egyptian children.

DETAILED DESCRIPTION:
Child's OHRQoL is assessed in terms of four main categories: oral symptoms as pain and discomfort, functional limitations as reduced masticatory efficiency due to malocclusion, emotional limitations as reduced self-esteem and social limitations as being teased by other children.

Deleterious Oral Habit is believed to be associated with emotional disturbances and orofacial dysfunction which will certainly affect child's OHRQoL.

Sucking habits, mouth breathing habits and tongue thrusting habits are found to be the most deleterious habits, especially in the selected age group of (5-7) years. It was found that these three deleterious habits are the most practiced habits among Egyptian children aging from 6-9 years (19.6%).

Up to the investigator's knowledge, there are very scanty studies investigating the effect of orofacial dysfunction on OHRQoL in children, only one of them was conducted on children practicing oral habits, but none of them was conducted on Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative Egyptian children aging from (5 - 7) years.
* Medically free children.
* Children whose families accept to participate in this study.

Exclusion Criteria:

* Children with untreated caries.
* Children with previous untreated dental trauma.
* Children with previous orthodontic treatment
* Children with upper respiratory disease
* Children having one or more of the following conditions: MIH, amelogenesis imperfecta, dentinogenesis imperfecta, hypodontia, dental fluorosis.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Egyptian children aging from 5 to 7 years old.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Orofacial dysfunction | Baseline: Child will be examined for once.
  Measured by Nordic Orofacial Test Screen. Measuring Unit: Scores (from 0 to 12) consists of two main parts: First part is NOT-S Interview and the second part is NOT-S Examination. Each part contains six domains as following (Appendix 2):
  • NOT-S Interview: I. Sensory function. II. Breathing. III. Habits. IV. Chewing and swallowing. V. Drooling. VI. Dry mouth.
  • NOT-S Examination:
  1. Face at rest.
  2. Nose breathing.
  3. Facial expression.
  4. Masticatory muscle and jaw function.
  5. Oral motor function.
  6. Speech

SECONDARY OUTCOMES:
Oral Health Related Quality of Life | Baseline: the questionnaire will be filled by child's caregiver for once.
  Measured by: Parental Caregiver Perciption Questionnaire and Family Impact Scale. Measuring Unit: Scores, For Parental-Caregiver Perception Questionnaire: from 0 to 32 For Family Impact scale : from 0 to 32.
  * Parental- Caregiver Perception Questionnaire consists of 4 sections:
    1. Oral symptoms domain (2 items).
    2. Functional limitation domain (2 items).
    3. Emotional well-being domain (2 items).
    4. Social well-being domain (2 items).
  * Family Impact Scale consists of 3 sections:
    1. Parental emotions domain (2 items).
    2. Parental / family activity domain (4 items).
    3. Family conflict domain (2 items).

CONTACTS AND LOCATIONS:
Overall Officials: Mennat Allah A.Elkareem, B.D.S, Principal Investigator — Fuculty of Dentistry, Ahram Canadian University
Locations (1):
- Postgraduate clinics in Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egyp, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leme MS, Souza Barbosa Td, Gaviao MB. Relationship among oral habits, orofacial function and oral health-related quality of life in children. Braz Oral Res. 2013 May-Jun;27(3):272-8. doi: 10.1590/S1806-83242013000300006. PMID 23739786
- [Background] Al-Riyami IA, Thomson WM, Al-Harthi LS. Testing the Arabic short form versions of the Parental-Caregivers Perceptions Questionnaire and the Family Impact Scale in Oman. Saudi Dent J. 2016 Jan;28(1):31-5. doi: 10.1016/j.sdentj.2015.08.001. Epub 2015 Nov 22. PMID 26792967
- [Background] Kumar S, Kroon J, Lalloo R, Johnson NW. Validity and reliability of short forms of parental-caregiver perception and family impact scale in a Telugu speaking population of India. Health Qual Life Outcomes. 2016 Mar 1;14:34. doi: 10.1186/s12955-016-0433-7. PMID 26932786
- [Background] Bakke M, Bergendal B, McAllister A, Sjogreen L, Asten P. Development and evaluation of a comprehensive screening for orofacial dysfunction. Swed Dent J. 2007;31(2):75-84. PMID 17695052
- [Derived] Abd-Elsabour MAAA, Hanafy RMH, Omar OM. Effect of self-perceived oral habits on orofacial dysfunction and oral health-related quality of life among a group of Egyptian children: a cohort study. Eur Arch Paediatr Dent. 2022 Dec;23(6):935-944. doi: 10.1007/s40368-022-00740-8. Epub 2022 Aug 24. PMID 36001236